CLINICAL TRIAL: NCT06956690
Title: A First-in-Human, Open-label, Phase 1/2 Clinical Trial to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of HMBD-501 in Patients With Advanced-Stage, Relapsed/Refractory HER3-Expressing Solid Tumors
Brief Title: A Phase 1/2 Clinical Trial to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of HMBD-501 in Patients With HER3-Expressing Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hummingbird Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMBD-501-101
Record Dates: First submitted 2025-04-24; First posted 2025-05-04 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Melanoma (Skin); Non Small Cell Lung Cancer; Breast Cancer
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HMBD-501 (Experimental): HMBD-501 intravenous injection once every 3 weeks; successive cohorts will receive escalating doses of HMBD-501 until the RP2D is reached
  Interventions: Biological: ENV-501

INTERVENTIONS:
Biological: ENV-501 — ENV-501 is a HER3-targeted antibody-drug conjugate (ADC) with a humanized monoclonal antibody (mAb) conjugated with a chemotherapeutic payload via a linker.

SUMMARY:
This study is a Phase 1/2, first-in-human, open-label, clinical trial to assess the safety, tolerability, pharmacokinetics and preliminary efficacy of HMBD-501 in patients with advanced-stage, relapsed and/or refractory human epidermal growth factor receptor 3 (HER3)-expressing solid tumors. The study consists of 2 phases: a dose escalation phase (Phase 1) and a dose expansion phase (Phase 2).

The primary objectives of Phase 1 are to characterize the overall safety and tolerability profile of increasing doses of HMBD-501 in patients with advanced-stage solid tumors and identify the recommended Phase 2 dose (RP2D) of ENV-501. During Phase 1, successive cohorts of patients will receive escalating doses of HMBD-501. The results of the dose escalation will determine the RP2D and dosing schedule of HMBD-501 to be administered in the Phase 2 part of the study. The primary objective of Phase 2 is to evaluate the preliminary clinical efficacy of HMBD-501 in dose expansion cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥ 40 kg.
* Willing and able to provide signed written informed consent before any study-related screening procedures are performed.
* Patients with histologically or cytologically confirmed diagnosis of advanced-stage or metastatic HER3+ solid tumors that are relapsed or refractory to or ineligible for standard therapy, or for whom no standard therapy is available; or the patient has documented their refusal of standard of care therapies. These include the following:

  1. Unresectable or metastatic cutaneous melanoma (HER3+)
  2. Locally advanced or metastatic mutated EGFR (mEGFR) NSCLC (HER3+)
  3. Unresectable, locally advanced or metastatic breast cancer
  4. Relapsed or refractory solid tumors, with documented HER3+ expression such as Pancreatic Ductal Adenocarcinoma (PDAC) and gastric cancers, may be allowed in the protocol following sponsor approval on a case-by -case basis.
* If molecular pathology report to confirm HER3+ status is not available, willingness to undergo fresh tumor biopsy for retrospective assessment of HER3+ status following enrollment..
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2.
* Contraceptive requirements:

  1. Women of childbearing potential (WOCBP) must use contraception from at least 28 days prior to study start, during the study, and for at least 6 months after the last dose of study drug.
  2. Males who are sexually active with partner(s) who are WOCBP must agree to use a male condom with spermicide beginning at study start, during the study and for at least 6 months after the last dose of study drug.
* Females must:

  1. Agree to not donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 6 months after the last dose of study drug.
  2. Agree to not breastfeed and do not plan to become pregnant during the study and for at least 6 months after the last dose of study drug.
* Males must:

  1. Agree to not donate sperm beginning at study start, during the study, and for at least 6 months after the last dose of study drug.
  2. Agree to not plan to father a child beginning at study start, during the study, and for at least 6 months after last dose of study drug.
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Any of the following treatment interventions within the specified time frame prior to study drug administration at study start:

  1. Any anti-tumor-directed drug therapy within 21 days or 5 times the elimination half-life (whichever is shorter).
  2. Treatment with investigational drugs within 21 days.
  3. Major surgery within 21 days.
  4. Radiation therapy ≤4 weeks or radiotherapy that included >30% of the bone marrow.
  5. Autologous or allogeneic stem cell transplantation or allogeneic tissue/organ transplant within 3 months.
  6. CYP3A4 strong inhibitor (including any prescription or non-prescription drugs or herbal supplements) ≤4 half-lives.
  7. CYP3A4 strong inducer ≤4 half-lives.
  8. OATP1B inhibitor (including any prescription or non-prescription drugs or herbal supplements) ≤4 half-lives.
* Prior treatment with a HER3-targeted ADC or any exatecan- or exatecan-derivative-conjugated ADC inhibitor as last line of therapy.
* Prior treatment with a topoisomerase I inhibitor as last line of therapy.
* Primary immune deficiency (e.g. congenital syndromes).
* Active and uncontrolled infections requiring intravenous antibiotic or antiviral treatment within 2 weeks prior to study start.
* Known/suspected hypersensitivity against ENV-501, human or humanized immunoglobulin Gs (IgGs), or their ingredients.
* History of noninfectious or drug-induced pneumonitis or interstitial lung disease (ILD).
* Known seropositivity (except after vaccination or confirmed cure for hepatitis) for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).
* Leptomeningeal disease, symptomatic or uncontrolled (active) brain metastasis (note: brain metastases not requiring steroids or anti-epileptic therapy are allowed if stable for ≥4 weeks prior to study start and patient is neurologically stable).
* Pregnant or WOCBP who have a positive b-human chorionic gonadotropin (HCG) test result at Screening or within 7 days prior to study start.
* Patients with second malignancies that are active (uncontrolled, metastatic) or requiring therapy.
* Patient who is an immediate family member (spouse, parent, child, or sibling; biological or legally adopted) of personnel directly affiliated with the study site or the Sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Phase 1 (Dose Escalation): Frequency of treatment-emergent adverse events | through study completion, an average of 6 months
Phase 2 (Dose Expansion): Objective Response Rate (ORR) | through study completion, an average of 6 months
  Objective Response is defined as Complete Response (CR) or Partial Response (PR) by investigator assessment, measured by revised Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
Phase 1 (Dose Escalation): Disease Control Rate (DCR) | through study completion, an average of 6 months
  DCR is defined as CR, PR, or Stable Disease (SD) by investigator assessment, measured by revised RECIST 1.1.
Phase 1 (Dose Escalation): Objective Response Rate (ORR) | through study completion, an average of 6 months
Phase 1 (Dose Escalation): maximum blood concentration (Cmax) after a single dose | At the end of Cycle 1 (each cycle is 21 days)
Phase 1 (Dose Escalation): time of maximum blood concentration (Tmax) after a single dose | At the end of Cycle 1 (each cycle is 21 days)
Phase 1 (Dose Escalation): absorption to time t (AUC0-t) after a single dose | At the end of Cycle 1 (each cycle is 21 days)
  AUC represents "area under the concentration-time curve" and measures the amount of drug that is present in the blood from the time of administration to a given time 't'
Phase 1 (Dose Escalation): absorption to end of the dosing period (AUC0-tau) after a single dose | At the end of Cycle 1 (each cycle is 21 days)
Phase 1 (Dose Escalation): total absorption (AUC0-infinity) after a single dose | At the end of Cycle 1 (each cycle is 21 days)
Phase 1 (Dose Escalation): drug half-life (t1/2) after a single dose | At the end of Cycle 1 (each cycle is 21 days)
Phase 1 (Dose Escalation): minimum blood concentration (Cmin) after a single dose | At the end of Cycle 1 (each cycle is 21 days)
Phase 1 (Dose Escalation): rate of clearance (CL) after a single dose | At the end of Cycle 1 (each cycle is 21 days)
Phase 1 (Dose Escalation): steady-state volume of distribution (Vss) after a single dose | At the end of Cycle 1 (each cycle is 21 days)
Phase 1 (Dose Escalation): Cmax at steady state | through study completion, an average of 6 months
Phase 1 (Dose Escalation): Tmax at steady state | through study completion, an average of 6 months
Phase 1 (Dose Escalation): AUC0-t at steady state | through study completion, an average of 6 months
Phase 1 (Dose Escalation):AUC0-tau at steady state | through study completion, an average of 6 months
Phase 1 (Dose Escalation): t1/2 at steady state | through study completion, an average of 6 months
Phase 1 (Dose Escalation): Cmin at steady state | through study completion, an average of 6 months
Phase 1 (Dose Escalation): accumulation ratio at steady state | through study completion, an average of 6 months
Phase 2 (Dose Expansion): Disease Control Rate (DCR) | through study completion, an average of 6 months
Phase 2 (Dose Expansion): Duration of Response (DoR) | through study completion, an average of 6 months
  A DoR event is defined as disease progression or death due to any cause in the subset of patients who achieved CR or PR on the study. DoR will be calculated from the date of first radiographic evidence of objective response by RECIST v1.1 to the date of progression, date of death, or date of last follow-up, whichever is the earliest.
Phase 2 (Dose Expansion): Progression-free Survival (PFS) | through study completion, an average of 6 months
  A PFS event is defined as disease progression or death due to any cause. PFS will be calculated from the date of treatment start to the date of progression, date of death, or date of last follow-up, whichever is the earliest.
Phase 2 (Dose Expansion): Frequency of treatment-emergent adverse events | through study completion, an average of 6 months
Phase 2 (Dose Expansion): Cmax at steady state | through study completion, an average of 6 months
Phase 2 (Dose Expansion): Cmin at steady state | through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Lancaster, M.D., Study Director — Endeavor Biomedicines
Locations (6):
- United States (4):
  - Research Site, La Jolla, California
  - Research Site, Indianapolis, Indiana
  - Research Site, Farmington Hills, Michigan
  - Research Site, Dallas, Texas
- Australia (2):
  - Research Site, Campbelltown, New South Wales
  - Research Site, Miranda, New South Wales

IPD SHARING:
Plan to Share IPD: No